CLINICAL TRIAL: NCT02780375
Title: Feasibility Study Testing Multi-panel Coding and Non-coding Transcriptional Responses as an Indicator of Individualised Responses to Radiation Effects in Radiation Therapy Patients
Brief Title: Feasibility Study Testing Transcriptional Responses as an Indicator of Individualised Responses to Radiation Effects
Acronym: RTGene
Status: Completed | Type: Observational
Sponsor: Institute of Cancer Research, United Kingdom (Other)
Collaborators: Public Health England (Other Government)
Responsible Party: Sponsor
Other Study IDs: CCR4553
Record Dates: First submitted 2016-05-13; First posted 2016-05-23 (Estimated); Last update posted 2018-10-31 (Actual); Status verified 2018-10

CONDITIONS: Cancer
Keywords: Transcriptional Responses; Radiation
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Blood donation during radiotherapy: Participants will be asked to donate a blood sample at 5 time points before and during their radiotherapy
  Interventions: Procedure: Blood donation during radiotherapy

INTERVENTIONS:
Procedure: Blood donation during radiotherapy — Participants will be asked to donate a blood sample at 5 time points before and during their radiotherapy

SUMMARY:
Peripheral blood samples will be taken with informed consent from radiotherapy patients undergoing standard radiotherapy at The Royal Marsden before and during treatment for breast, lung, gastrointestinal and genitourinary tumours. Responses from panels of up to 800 coding and non-coding RNAs will be assessed in the samples using the nCounter system. Candidate genes identified by Public Health England, Columbia University and/or in the literature as being specific to radiation responses will be included, together with genes relevant to systemic inflammatory responses, to identify transcriptional responses for a range of doses and exposures on an inter-individual basis. Data will be analysed using existing and new statistical tools focused on count data modelling. The intended outcome is identification of a radiation specific panel of genes to inform individual radiation responses and if the results are favourable, a large scale follow up to this proposed pilot is expected in due course.

DETAILED DESCRIPTION:
Biological markers of radiation exposure play a crucial role in the triage of suspected exposed persons following a radiation accident or incident. They can also estimate individual doses that enable assessment of late radiation effects in affected individuals. In recent years the gene expression assay has been shown to be a sensitive biological marker of radiation exposure with the potential to be used for truly individualised dosimetry. The possibility for this gene expression assay to be used in a large scale mass-casualty scenario has been proposed and tested in a recent intercomparison exercise. Classic cytogenetic techniques, and in particular the gold standard dicentric assay, have two main disadvantages: (1) lack of high-throughput and (2) delays of several days between blood sampling and the availability of results. Although more work needs to be done to further assess its suitability for triage purposes, it is clear that gene expression analysis in blood samples can provide valuable information, as there is a window of time (i.e. 12-48 hours) following radiation exposure where specific radiation-responsive genes have linear dose responses (0-5 Gy). Most work to date has focused on developing sensitive assays for studying gene expression modifications using state of the art technology, i.e. multiplex quantitative, digital polymerase chain reaction (qPCR) and molecular counting systems.

At Public Health England (PHE), recently established technology allows direct counting of nucleic acid molecules (DNA, mRNA, miRNA and lncRNA) without the need for enzymatic reaction or amplification steps hence reducing time for data collection. The system offers multiplexing capacity comparable to microarrays but with greater precision and sensitivity. Another unique advantage of this technology is that there is no need for long, time consuming bioinformatic analyses as the results are obtained as counted number of events. This new gene expression analysis technique has been assessed for radiation biodosimetry applications with promising results. Furthermore, gene expression has shown a high degree of promise as a marker for late effects of radiation, for instance normal tissue reactions following curative radiotherapy for breast cancer. Clinical data suggest that systemic inflammatory responses plays a critical role in the progression of radiation effects: for instance, the neutrophil-to-lymphocyte ratio represents a marker of systemic inflammation pre-treatment and is an independent prognostic factor useful for individual risk assessment in breast cancer patients undergoing radiotherapy. Genes relevant to inflammatory responses are thus interesting candidates for further investigation. Linearity of the transcriptional dose-response for specific radiation-responsive genes in ex vivo exposed human blood samples has recently been demonstrated for the first time, and inter-individual variability in the response after low doses and high doses exposures has been newly assessed. The logical next stage for biological development of the gene expression assay is to validate these new techniques with human blood samples exposed to radiation in vivo.

The use of samples from patients undergoing radiotherapy for validation of techniques has been gaining popularity in recent years. Sophisticated treatment planning for clinical radiotherapy leads to very accurate individual dose calculations that allow for validation of biological estimates of dose. The range of standard radiotherapy schedules chosen for inclusion in this study will provide a wide range of doses for assessment of the gene expression assay alone and in combination with the other cytogenetic assays, to simulate a range of potential exposure scenarios.

Peripheral blood samples will be taken with informed consent from patients undergoing standard radiotherapy before and during treatment for breast, lung, gastrointestinal and genitourinary tumours. Responses from panels of up to 800 coding and non-coding RNAs will be assessed in the samples using the nCounter system. Candidate genes identified by PHE, Columbia and/or in the literature as being specific to radiation responses will be included, together with genes relevant to systemic inflammatory responses, to identify transcriptional responses for a range of doses and exposures on an inter-individual basis. Data will be analysed using existing and new statistical tools focused on count data modelling. The intended outcome is identification of a radiation specific panel of genes to inform individual radiation responses and if the results are favourable, a large scale follow up to this proposed pilot is expected in due course.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Requirement for external beam radiotherapy for breast, lung, gastrointestinal or genitourinary tumours
* Written informed consent

Exclusion Criteria:

* Previous radiotherapy
* Concurrent chemotherapy or chemotherapy preceding radiotherapy by less than 4 weeks
* Concurrent hormone therapy or hormone therapy preceding radiotherapy by less than 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing radiotherapy for cancer
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2016-09-12 (Actual); Primary Completion 2018-07-17 (Actual); Study Completion 2018-07-17 (Actual)

PRIMARY OUTCOMES:
Transcriptional responses as measured by nCounter molecular profiling as biomarker of individual radiation exposure | 3 months after all volunteers have finished radiotherapy and donated blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Navita Somaiah, Principal Investigator — Institute of Cancer Research, United Kingdom
Locations (1):
- The Royal Marsden, Sutton, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lloyd, D.C. and A.A. Edwards, Biological dosimetry after radiation accidents. In: G. Obe et al.,(eds). Chromosomal Aberrations. Springer-Verlag, Berlin, Heidelberg. 1990.
- [Background] Maznik, N.A., et al., Chromosomal dosimetry for some groups of evacuees from Prypiat and Ukrainian liquidators at Chernobyl. Radiation Protection Dosimetry, 1997. 74(1-2): p. 5-11.
- [Background] Kabacik S, Mackay A, Tamber N, Manning G, Finnon P, Paillier F, Ashworth A, Bouffler S, Badie C. Gene expression following ionising radiation: identification of biomarkers for dose estimation and prediction of individual response. Int J Radiat Biol. 2011 Feb;87(2):115-29. doi: 10.3109/09553002.2010.519424. Epub 2010 Nov 10. PMID 21067298
- [Background] Manning G, Kabacik S, Finnon P, Bouffler S, Badie C. High and low dose responses of transcriptional biomarkers in ex vivo X-irradiated human blood. Int J Radiat Biol. 2013 Jul;89(7):512-22. doi: 10.3109/09553002.2013.769694. Epub 2013 Feb 27. PMID 23362884
- [Background] Kabacik S, Ortega-Molina A, Efeyan A, Finnon P, Bouffler S, Serrano M, Badie C. A minimally invasive assay for individual assessment of the ATM/CHEK2/p53 pathway activity. Cell Cycle. 2011 Apr 1;10(7):1152-61. doi: 10.4161/cc.10.7.15231. Epub 2011 Apr 1. PMID 21389785
- [Background] Badie C, Kabacik S, Balagurunathan Y, Bernard N, Brengues M, Faggioni G, Greither R, Lista F, Peinnequin A, Poyot T, Herodin F, Missel A, Terbrueggen B, Zenhausern F, Rothkamm K, Meineke V, Braselmann H, Beinke C, Abend M. Laboratory intercomparison of gene expression assays. Radiat Res. 2013 Aug;180(2):138-48. doi: 10.1667/RR3236.1. Epub 2013 Jul 25. PMID 23886340
- [Background] Ainsbury EA, Bakhanova E, Barquinero JF, Brai M, Chumak V, Correcher V, Darroudi F, Fattibene P, Gruel G, Guclu I, Horn S, Jaworska A, Kulka U, Lindholm C, Lloyd D, Longo A, Marrale M, Monteiro Gil O, Oestreicher U, Pajic J, Rakic B, Romm H, Trompier F, Veronese I, Voisin P, Vral A, Whitehouse CA, Wieser A, Woda C, Wojcik A, Rothkamm K. Review of retrospective dosimetry techniques for external ionising radiation exposures. Radiat Prot Dosimetry. 2011 Nov;147(4):573-92. doi: 10.1093/rpd/ncq499. Epub 2010 Dec 23. PMID 21183550
- [Background] Kabacik S, Manning G, Raffy C, Bouffler S, Badie C. Time, dose and ataxia telangiectasia mutated (ATM) status dependency of coding and noncoding RNA expression after ionizing radiation exposure. Radiat Res. 2015 Mar;183(3):325-37. doi: 10.1667/RR13876.1. Epub 2015 Mar 4. PMID 25738893
- [Background] Manning, G., et al., Assessing a new gene expression analysis technique for radiation biodosimetry applications. Radiation Measurements, 2011. 46(9): p. 1014-1018.
- [Background] Finnon P, Kabacik S, MacKay A, Raffy C, A'Hern R, Owen R, Badie C, Yarnold J, Bouffler S. Correlation of in vitro lymphocyte radiosensitivity and gene expression with late normal tissue reactions following curative radiotherapy for breast cancer. Radiother Oncol. 2012 Dec;105(3):329-36. doi: 10.1016/j.radonc.2012.10.007. Epub 2012 Nov 15. PMID 23157981
- [Background] Krenn-Pilko S, Langsenlehner U, Stojakovic T, Pichler M, Gerger A, Kapp KS, Langsenlehner T. The elevated preoperative derived neutrophil-to-lymphocyte ratio predicts poor clinical outcome in breast cancer patients. Tumour Biol. 2016 Jan;37(1):361-8. doi: 10.1007/s13277-015-3805-4. Epub 2015 Jul 29. PMID 26219894
- [Background] Chua ML, Horn S, Somaiah N, Davies S, Gothard L, A'Hern R, Yarnold J, Rothkamm K. DNA double-strand break repair and induction of apoptosis in ex vivo irradiated blood lymphocytes in relation to late normal tissue reactions following breast radiotherapy. Radiat Environ Biophys. 2014 May;53(2):355-64. doi: 10.1007/s00411-014-0531-z. Epub 2014 Mar 13. PMID 24622963
- [Background] Chua ML, Somaiah N, A'Hern R, Davies S, Gothard L, Yarnold J, Rothkamm K. Residual DNA and chromosomal damage in ex vivo irradiated blood lymphocytes correlated with late normal tissue response to breast radiotherapy. Radiother Oncol. 2011 Jun;99(3):362-6. doi: 10.1016/j.radonc.2011.05.071. Epub 2011 Jun 23. PMID 21704405
- [Background] Chua ML, Somaiah N, Bourne S, Daley F, A'hern R, Nuta O, Davies S, Herskind C, Pearson A, Warrington J, Helyer S, Owen R, Yarnold J, Rothkamm K. Inter-individual and inter-cell type variation in residual DNA damage after in vivo irradiation of human skin. Radiother Oncol. 2011 May;99(2):225-30. doi: 10.1016/j.radonc.2011.04.009. Epub 2011 May 26. PMID 21620495
- [Background] Prise KM, O'Sullivan JM. Radiation-induced bystander signalling in cancer therapy. Nat Rev Cancer. 2009 May;9(5):351-60. doi: 10.1038/nrc2603. Epub 2009 Apr 20. PMID 19377507